CLINICAL TRIAL: NCT07357155
Title: An Observational Study of Oral and Salivary Biomarkers Associated With Stroke
Brief Title: Oral and Salivary Biomarkers Associated With Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Center (CHU) of Constantine, Algeria (Other Government)
Responsible Party: Principal Investigator, Abdeldjalil ZITOUNI, Principal Investigator, University Hospital Center (CHU) of Constantine, Algeria
Other Study IDs: CHU-STROKE-001
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: Stroke; Oral health; Salivary biomarkers; Cerebrovascular disease; Observational study
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Unstimulated saliva samples collected for the analysis of inflammatory and biochemical biomarkers. No genetic or DNA analysis will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke group: Patients diagnosed with stroke.
- Healthy control group: Healthy participants without a history of stroke.

SUMMARY:
This observational study aims to explore the association between oral and salivary biomarkers and stroke. The study will include adult participants diagnosed with stroke and will analyze clinical, oral, and salivary parameters. The objective is to improve understanding of potential links between oral health, salivary biomarkers, and cerebrovascular disease. No experimental intervention will be performed.

DETAILED DESCRIPTION:
Stroke is a major cause of morbidity and mortality worldwide. Growing scientific evidence suggests that oral health and salivary biomarkers may reflect systemic inflammatory and vascular conditions.

This observational study is designed to evaluate associations between oral clinical findings, salivary biomarkers, and stroke. Participants with a confirmed diagnosis of stroke will be enrolled. Data collection will include demographic information, medical history, oral examination findings, and salivary samples.

Analyses will focus on identifying correlations between oral and salivary parameters and clinical characteristics of stroke. This study does not involve any therapeutic intervention or experimental treatment. The findings may contribute to a better understanding of the oral-systemic relationship in cerebrovascular diseases and support future preventive strategies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 90 years.
* Patients diagnosed with stroke (ischemic or hemorrhagic) confirmed by clinical and imaging criteria for the stroke group.
* Healthy volunteers without a history of stroke or cerebrovascular disease for the control group.
* Ability to provide written informed consent.

Exclusion Criteria:

* inflammatory disease at the time of sampling.
* Chronic autoimmune or malignant disease.
* Recent major surgery or trauma within the last 3 months.
* Pregnancy or breastfeeding.
* Inability or refusal to provide saliva samples.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from multiple regions within Algeria, reflecting a diverse national population.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Differences in salivary inflammatory biomarker profiles between stroke patients and healthy controls. | Single time-point assessment at enrollment
  Assessment of salivary inflammatory and neuroendocrine biomarkers, including salivary cortisol and selected inflammatory cytokines (e.g., IL-6 and/or hs-CRP), to identify biomarker patterns associated with stroke.

SECONDARY OUTCOMES:
Exploratory association between oral microbiota profiles and stroke status | Single time-point assessment at enrollment
  Exploratory analysis of the association between oral microbiota profiles and stroke status using saliva or oral swab samples. The analysis aims to identify bacterial profiles potentially associated with stroke and oral-systemic interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Abdeldjalil Zitouni, DDS, Principal Investigator — Independent Researcher, Constantine, Algeria
Locations (1):
- Private Dental Clinic, Constantine, Constantine, Algeria

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality considerations.

REFERENCES:
- [Background] Miyatani F, et al. Collagen-binding activity of Streptococcus mutans and cerebral microbleeds. Stroke. 2015.